CLINICAL TRIAL: NCT04709393
Title: The Effects of FRAX+SARC-F Questionnaire Pre-screening on Promoting Public Awareness of Fragility Fracture and Fall Prevention Among Community-dwelling Older Adults
Brief Title: Effects of FRAX+SARC-F Pre-screening on Preventing Fragility Fracture and Fall in Community-dwelling Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020.609-T
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Age Related Osteoporosis; Fall
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-screening (Experimental): Receiving FRAX+SARC-F questionnaire pre-screening results on estimated fracture risk
  Interventions: Other: FRAX+SARC-F questionnaire pre-screening
- Control (No Intervention): Not receiving FRAX+SARC-F questionnaire pre-screening preliminary results on estimated fracture risk

INTERVENTIONS:
Other: FRAX+SARC-F questionnaire pre-screening — Pre-screening group participants will receive the FRAX+SARC-F questionnaire pre-screening and be notified of the preliminary estimation of their future hip fracture risk before being invited to our DXA screening and fall-risk assessment.
  Arms: Pre-screening

SUMMARY:
Hip fragility fractures are a major threat to functional independence in older adults locally and globally. In Hong Kong, the prevalence of osteoporosis and osteopenia in people aged >50 years were reported to be as high as 37% and 52%, respectively. The major challenge in fragility fracture prevention is that fragility fracture is caused by the combination of osteoporosis and propensity to fall, and both of these conditions are multifactorial. Ample evidence shows that fall risks can be reduced by well-designed exercises, and osteoporosis can be effectively diagnosed by Dual-energy X-ray Absorptiometry imaging (DXA) and treated with anti-osteoporosis medication. Lifestyle modifications e.g. diet, optimal physical activity, environmental safety can also help to prevent falls or improve bone health. The brief Fracture Risk Assessment Tool (FRAX) and SARC-F provide a low cost of prescreening for fracture risk and sarcopenia, respectively. Using SARC-F in conjunction with FRAX has increased sensitivity for hip fracture risk prediction. FRAX+SARC-F may help increase the public awareness of osteoporosis and get the at-risk group to receive diagnostic tests and be treated. This model should fit in well with the coming District Health Centres across Hong Kong.

DETAILED DESCRIPTION:
Participants will be randomly assigned to either the pre-screening or control group in a 1:1 ratio. Independent personnel not involved in data collection or intervention will perform and conceal the randomization using an online data server. Research assistants who are blinded to the group allocation will conduct all the baseline assessments and subsequent event surveillance. All data will also be entered and checked by the blinded research assistants. All procedures concur with the Declaration of Helsinki (2013).

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 65 years
* living in the community

Exclusion Criteria:

• cannot follow the instruction

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2956 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
proportions of participants diagnosed with osteoporosis in the FRAX+SARC-F pre-screening and control groups. | within 1-6 months
  proportions of participants diagnosed with osteoporosis in the FRAX+SARC-F pre-screening and control groups.

SECONDARY OUTCOMES:
Rate of receiving osteoporosis screening | 6-12 months
  Number of participants receiving osteoporosis screening in the arms
rate of receiving fall risk assessment | 6-12 months
  Number of participants receiving fall risk assessment in the arms
rate of receiving anti-osteoporosis intervention | 6-12 months
  Number of participants receiving anti-osteoporosis intervention in the arms
rate of receiving fall prevention intervention | 6-12 months
  Number of participants receiving fall prevention intervention in the arms
subsequent fall rate | 12 months
  Number of participants having subsequent fall in the arms
subsequent fracture rate | 12 months
  Number of participants having subsequent fracture in the arms

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kwok, Principal Investigator — The Chinese University of Hong Kong Jockey Club Centre for Osteoporosis Care and Control
Locations (1):
- The Chinese University of Hong Kong Jockey Club Centre for Osteoporosis Care and Control, Hong Kong, Hong Kong